CLINICAL TRIAL: NCT06884293
Title: A Multicenter, Randomized, Open-label Phase III Study to Compare the Efficacy and Safety of IBI362 and Semaglutide in Chinese Overweight or Obese Subjects With Metabolic Dysfunction-associated Fatty Liver Disease (GLORY-3)
Brief Title: A Study Comparing IBI362 vs Semaglutide in Chinese Overweight or Obese Adults With Metabolic Dysfunction-associated Fatty Liver Disease （MAFLD）
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI362B303
Record Dates: First submitted 2025-03-11; First posted 2025-03-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Overweight; Metabolic Dysfunction-associated Fatty Liver Disease (MAFLD)
MeSH Terms: conditions — Overweight | interventions — mazdutide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Active Comparator)
  Interventions: Drug: semaglutide
- IBI362 (Experimental)
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: IBI362 — Once-weekly injections of gradually increased doses of IBI362, subcutaneously (SC): starting dose is 2.0 mg, after 4 weeks of administration, increase to 4.0 mg; After another 4 weeks, increase to 6mg; After another 4 weeks, increase to the maximum dose 9mg for 36 weeks
  Arms: IBI362
Drug: semaglutide — Once-weekly injections of gradually increased doses, subcutaneously (SC): starting dose is 0.25 mg, after 4 weeks of administration, increase to 0.5 mg; After another 4 weeks, increase to 1mg; After another 4 weeks, increase to 1.7mg; After another 4 weeks, increase to the maximum 2.5mg for 32 weeks
  Arms: Semaglutide

SUMMARY:
This is a multicenter, randomized, open-label Phase 3 clinical study comparing the efficacy and safety of IBI362 9 mg QW versus Semaglutide 2.4 mg QW in overweight or obese (BMI≥27kg/m2) MAFLD subjects. Subjects will be randomly assigned to IBI362 9 mg and Semaglutide 2.4 mg groups. All study treatment will be administered once-weekly and subcutaneously. The entire trial cycle includes a 4-week screening period, a 48-week open-label treatment period, and a 12-week drug withdrawal safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older at the time of signing informed consent
2. diagnosed as MAFLD according to the Chinese Guideline for the prevention and treatment of metabolic dysfunction-associated (non-alcoholic) fatty liver disease (Version 2024)
3. liver fat content ≥8% measured by MRI-PDFF
4. BMI≥27 kg/m2
5. Weight change ≤5% within 3 months before screening
6. HbA1c≤10%

Exclusion Criteria:

1. Subjects who the investigator thinks may be allergic to the components in the study drug or similar drugs
2. Used drugs or alternative therapies with weight loss effects within 3 months before screening, including but not limited to: GLP-1 receptor agonists, orlistat, phenylpropanolamine, chlorpheniramine, phentermine etc.
3. Received chronic (>2 weeks) systemic glucocorticoid treatment within 3 months before screening (excluding topical, intraocular, intranasal, and inhaled administration)
4. Previous diagnosis of type 1 diabetes (including adult latent autoimmune diabetes)
5. Active or untreated malignant tumors within 5 years before screening, or patients are in remission of clinical malignant tumors (except patients with skin basal cell carcinoma and squamous cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or papillary thyroid carcinoma who have no recurrence after surgery)
6. Mental illness existed in the past or at the time of screening, and the researcher thinks it is not suitable to participate in this study
7. Pregnant or lactating women, or men or women who are fertile and unwilling to use contraception throughout the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
percentage change in body weight from baseline | at Week 48
percentage change in liver fat content from baseline measured by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) | at Week 48

SECONDARY OUTCOMES:
percentage change in liver fat content from baseline measured by MRI-PDFF | at Week 8, 16, and 24
Absolute value change in liver fat content from baseline measured by MRI-PDFF | at Week 8, 16, 24, and 48
Proportion of subjects with weight loss >10% from baseline and liver fat content <5% | at week 48
percentage change in body weight from baseline | at week 24
Changes in systolic blood pressure and diastolic blood pressure from baseline | at week 48
percentage changes in total cholesterol,triglyceride (TG), non-High Density Lipoprotein Cholesterol (non-HDL-C), Low Density Lipoprotein Cholesterol (LDL-C), HDL-C (High Density Lipoprotein Cholesterol) from baseline | at week 48
Changes in serum uric acid from baseline | at week 48
Changes in hemoglobin A1c (HbA1c) from baseline | at week 48
Changes in Homeostasis Model Assessment 2-B (HOMA2-B) from baseline | at week 48
Changes in Homeostasis Model Assessment 2-IR (HOMA2-IR) from baseline | at week 48
Changes of scores in 36-item Short-Form Health Survey version 2(SF-36v2) questionnaire from baseline | at week 48
  Using norm-based scoring (NBS)，each subscale has a different maximum and minimum score, with higher scores reflecting better levels of functioning
Changes of scores in The Impact of Weight on Quality of Life-Lite Clinical Trials Version(IWQoL-Lite-CT) questionnaire from baseline | at week 48
  Total score ranging from 0 to 100, with higher scores reflecting better levels of functioning

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Guo, M.D, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No